CLINICAL TRIAL: NCT06795841
Title: Photobiomodulation Therapy Versus Integrated Myofascial Release Therapy Techniques In Patients With Moderate COVID 19 Inside Intensive Care Unit, With a Complementary Home Telerehabilitation
Brief Title: Photobiomodulation Therapy Versus Integrated Myofascial Release Therapy Techniques In Patients With COVID-19 With Follow-Up Telerehabilitation
Acronym: PBM in COVID19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sherin Hassan Mohammed Mehani, Professor at Faculty of Physical Therapy - Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FBTBSUREC/2052020; FBTBSUREC/2052020 (Registry Identifier: Faculty of Physical Therapy = Beni-Suef University)
Record Dates: First submitted 2025-01-20; First posted 2025-01-28 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: COVID 19 Disease
Keywords: COVID19; Photobiomodulation; Myofascial release
MeSH Terms: conditions — COVID-19 | interventions — Low-Level Light Therapy; Myofascial Release Therapy; Telerehabilitation

STUDY DESIGN:
Intervention Model Description: The intervention group (A) consisted of 34 patients (men and women) who received medical treatment, traditional physiotherapy, and low-level laser therapy; the intervention group (B) consisted of 34 patients ( men and women) who received medical treatment and traditional physiotherapy and myofascial release techniques; and the control group (C) consisted of 34 patients ( men and women ) who received medical treatment and traditional physiotherapy only.After discharge all patients received home multidimension telerehabilitation program for 3 month.
Who Masked: Outcomes Assessor
Masking Description: Data analyzer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Photobiomodulation therapy (Experimental): Photobiomodulation therapy :Red laser wavelength (630-660 nm), Average power: 50-100 Mw, Dose: 6-10 J/cm2• Area 2-3 minutes/cm2, Sessions: twice -daily, acupuncture Laser Positions: transcutaneous laser therapy
  Interventions: Radiation: Photobiomodulation; Other: telerehabilitation
- Myofascial release therapy (Experimental): Myofascial release therapy A- Suboccipital release technique B- anterior cervical myofascial release C- Anterior thoracic and sternal myofascial release D- diaphragmatic dome release technique in addition to traditional physical therapy program
  Interventions: Procedure: Myofascial release therapy; Other: telerehabilitation
- traditional physical therapy program (Experimental): included traditional chest physiotherapy (postural drainage, percussion and shaking), stretching exercise for ( strencliedo mastoid ,scalene muscle ,pectorals major and minor ,hamstring and calf muscles )
  Interventions: Device: traditional chest physiotherapy; Other: telerehabilitation

INTERVENTIONS:
Radiation: Photobiomodulation — It was applied for upper respiratory tract over tonsils, trachea, and main bronchi (bilaterally parasternal at the level of angle of Lewis), upper and lower lung, and at cubital vein
  Arms: Photobiomodulation therapy
Procedure: Myofascial release therapy — technique was applied from supine position, with both hands cupping both diaphragmatic domes
  Arms: Myofascial release therapy
Device: traditional chest physiotherapy — included traditional chest physiotherapy (postural drainage, percussion and shaking), stretching exercise
  Arms: traditional physical therapy program
Other: telerehabilitation — Following ICU discharge, all patients participated in a 12-week structured home multidimensional telerehabilitation program delivered via videoconferencing (Zoom or Microsoft Teams) under the remote supervision of a physiotherapist. Sessions were conducted three times per week and incorporated patient education, breathing exercises, inspiratory muscle training (30 -50% MIP), strengthening of upper and lower limb muscle groups (50- 70 % 1RM), aerobic training (40- 60% HRR), and trunk control activities. Safety monitoring was emphasized throughout, with patients instructed to use a pulse oximeter before, during, and after each session. Adherence was assessed by session attendance, exercise diaries, and weekly therapist follow-up

SUMMARY:
Objective: To compare low-level laser therapy and myofascial release in reducing inflammation and functional recovery in critically ill COVID-19 patients with 3-month home-based telerehabilitation assessment.

Participants: One hundred two COVID-19 patients aged 45-60 years randomized into three groups: low-level laser therapy (n=34), myofascial release (n=34), and control (n=34).

Intervention: Intensive care unit-based low-level laser therapy, myofascial release, or standard physiotherapy with medical treatment. Following discharge, all participants received 12 weeks of multidimensional home-based telerehabilitation incorporating patient education, breathing exercises, inspiratory muscle training, limb strengthening, aerobic training, and trunk control.

Outcomes: Primary outcomes were ferritin and D-dimer levels. Secondary outcomes included C-reactive protein, interleukin-6, white blood cell counts, maximum inspiratory pressure, six-minute walk test, bilateral knee strength, dyspnea perception, fatigue severity, and oxygen saturation. All measured at baseline, discharge, and 3 months. Intensive care unit length of stay and physiotherapy sessions measured at discharge.

DETAILED DESCRIPTION:
One hundred-two COVID 19 patients (56 men and 46 women) aged 45-60 years were recruited from the Al Kasr Al Ainy teaching hospitals ICUs. All patients were informed of the study, risks, and expected benefits before signing the informed consent form. The low-level laser therapy group (LLLT) consisted of 34 patients, who received low-level laser therapy, traditional physiotherapy, medical treatment and the myofascial release group (MR) consisted of 34 patients, who received myofascial release techniques, traditional physiotherapy, and medical treatment; and the control group (C) consisted of 34 patients, who received traditional physiotherapy and medical treatment only. After discharge all patients received home multidimension telerehabilitation program.

The eligibility criteria were as follows: (I) Patients aged from 45 to 60 years old, (II) Diagnosed by CT or PCR as positive COVID 19, (III) Moderate cases of COVID-19 (According to CO-RA DS Scale).22 (IV) on low flow rate oxygen supply Exclusion criteria were (I) patients on Invasive Mechanical Ventilation, (II) Hemodynamically Unstable with inotropic support; (III) Septic Shock; (IV) ICU admission less than 24 h.

(V) physician termination of physiotherapy; and (VI) fever with causes other than chest infection, (VII) severe electrolyte imbalance, acute venous thromboembolism without therapeutic anticoagulation for over 48 h, (VIII) Unstable Atrial fibrillation, or severe tachycardia compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* The eligibility criteria were as follows:
* Patients aged from 45 to 60 years old.
* Diagnosed by CT or PCR as positive COVID 19.
* Moderate cases of COVID-19(According to CO-RADS Scale).
* On low flow rate oxygen supply

Exclusion Criteria:

* Patients on Invasive Mechanical Ventilation
* Hemodynamically Unstable with inotropic support
* Septic Shock
* ICU admission less than 24 h
* physician termination of physiotherapy;
* Fever with causes other than chest infection.
* Severe electrolyte imbalance
* Acute Venous Thromboembolism (VTE) without therapeutic anticoagulation for over 48 hours,
* Unstable Atrial fibrillation , or Severe Tachycardia compared to baseline.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Lab Investigations | at baseline and at discharge from ICU up to 14 days and at 3 month of discharge
  (1) ferritin
lab investigation | at baseline and at icu discharge up to 14 days and at 3 months of discharge
  2. D-dimer

SECONDARY OUTCOMES:
lab analysis | at baseline and at ICU discharge up to 14 days and at 3 months of discharge
  (3) CRP
lab analysis | at baseline and at icu discharge up to 14 days and at 3 months of discharge
  (4) Interleukin-6
lab analysis | at baseline and at icu discharge up to 14 days and at 3 months of discharge
  (5) white blood cell counts.
Maximum inspiratory pressure | at baseline and at icu discharge upto 14 days and at 3 months of discharge
  Maximum inspiratory pressure
Six-minute walk test | at baseline and at ICU discharge up to 14 days and at 3 months of discharge
  The 6-minute walk test (6-MWT) was conducted in the intensive care unit under the supervision
Ease of breathing | at baseline and at ICU discharge up to 14 days and at 3 months of discharge
  It was assessed using visual analogue scale: Zero represented deep, comfortable breathing; 10 represented inability to breathe deeply. Scores were recorded on a graduated ruler
Dyspnea perception | at baseline and at ICU discharge, up to 14 days and at 3 months of discharge
  It was assessed during a six-minute walking test: modified Borg scale (0-10) assessed dyspnea: zero = no dyspnea; 10 = maximum dyspnea ever experienced
Percentage of oxygen saturation | at baseline and at ICU discharge up to 14 days and at 3 months of discharge
  portable intra-hospital patient monitor measured hemoglobin oxygen saturation in arterial blood.
Icu length of stay | at ICU discharge up to 2weeks
fatigue | at baseline and at ICU discharge up to 14 days and at 3 months of discharge
  The Fatigue Severity Scale:Nine-item scale with 7-point Likert responses (1=strongly disagree to 7=strongly agree). Total score represents arithmetic mean of item responses.
Lower limbs strength | at baseline and at ICU discharge upto 14 days and at 3 months of discharge
  Quadriceps strength

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Ibrahim Mahmoud, Lecturer, Principal Investigator — Faculty of Physical Therapy - Beni-Suef University
Locations (1):
- Faculty of Physical Therapy , Beni-Suef University, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Yes
IPD could be shared in the form of study protocol , full details about study procedure and summary about the results . The sharing is available through the study principal investigator ; Prof. Sherin Mehani for about 12 months after publishing the paper.
Supporting Information: Study Protocol
Time Frame: The sharing is available through the study principal investigator ; Prof. Sherin Mehani for about 12 months after publishing the paper.
Access Criteria: All of the interested readers could access the needed IPD and supportive information upon request through E- mail sherinhassin@yahoo.com
URL: https://www.researchgate.net/profile/Mehani-Sherin

REFERENCES:
- [Background] Azadeh SS, Esmaeeli Djavid G, Nobari S, Keshmiri Neghab H, Rezvan M. Light-Based Therapy: Novel Approach to Treat COVID-19. Tanaffos. 2023 Mar;22(3):279-289. PMID 38638386